CLINICAL TRIAL: NCT05712070
Title: Impact of Smart Watch Mobile Application on Risk Treatment of CardioVascular Disease
Brief Title: Mobile Application for Cardiovascular Risk Treatment
Acronym: iSMART-CV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Soo-Jin Kang, MD., PhD., Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2023-0003
Record Dates: First submitted 2023-01-26; First posted 2023-02-03 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-01

CONDITIONS: Hypertension; Hyperlipidemias; Chronic Disease; Lifestyle Risk Reduction
Keywords: smart healthcare
MeSH Terms: conditions — Hypertension; Hyperlipidemias; Chronic Disease; Risk Reduction Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- smart group (Experimental): Smartphone App-based healthcare
  Interventions: Behavioral: App-guided lifestyle modification
- control group (Active Comparator): a book-based self-education
  Interventions: Behavioral: A book-based self-education of lifestyle modification

INTERVENTIONS:
Behavioral: App-guided lifestyle modification — Smart watch and smartphone application-based life style modification for 12 weeks
  Arms: smart group
Behavioral: A book-based self-education of lifestyle modification — A take-home book-based self-education for lifestyle modification
  Arms: control group

SUMMARY:
This study is a randomized, open-label clinical trial to validate the efficacy and safety of smartphone app-guided life style modification for the management of hypertension and hyperlipidemia.

DETAILED DESCRIPTION:
The aim of the study is to verify the blood pressure (BP) reduction and lipid-lowering effect of ICT-based healthcare program (intervention) vs. conventional strategy (control). Health insurance subscribers (KYOBO Life Insurance Co., Ltd.) who are aged 20-54 years, and have a recent record of an office BP ≥140/90 mmHg or serum LDL-cholesterol ≥130 mg/dl will be recruited. Among them, android smartphone users with no use of anti-hypertensive or lipid-lowering drugs for ≥3 months prior to screening will be referred to physicians in Asan Medical Center, and 24-hour ambulatory BP monitoring and serum LDL-cholesterol will be checked for screening. Finally, the patients who have a diagnosis of essential hypertension (24-hour ambulatory systolic BP 130-159 mmHg) or hyperlipidemia (LDL-cholesterol ≥130 mg/dl), and are considered appropriate to be managed with non-pharmacological lifestyle modification for 12 weeks will be eligible for enrollment.

The patients with 24-hour ambulatory systolic BP 130-159 mmHg and serum LDL-cholesterol <130 mg/dl were classified as [Category 1]. [Category 2] includes the patients with 24-hour ambulatory systolic BP <130 mmHg and serum LDL-cholesterol ≥130 mg/dl. The patients with 24-hour ambulatory systolic BP 130-159 mmHg and serum LDL-cholesterol ≥130 mg/dl are included in [Category 3]. The subjects in each category will be randomly allocated into the intervention and control groups as a ratio 1:1.

All participants will respond a baseline questionnaire about health habits, health behavior patterns and quality of life, diet, exercise, etc. They are provided with details on lifestyle modifications, as recommended by the Korean Society of Hypertension and/or the Korean society of lipid & atherosclerosis. The patients in the intervention group will wear a smart watch (Galaxy watch4, Samsung Electronics Co., Ltd.) collecting their physical data (BP, heart rate, activity, fitness, etc.), and will use the smartphone application (Second Wind, Medi Plus Solution Co., Ltd.) that provides the personalized healthcare services for lifestyle modification in chronic disease (nutrition, activities & exercise, weight & BP control, sleep, stress, medication, smoking cessation), health education and online consulting. In the control group, a take-home book about chronic illness will be given for self-education.

At 12-week follow-up, 24-hour ambulatory BP monitoring and serum LDL-cholesterol measurement will be repeatedly done. The primary endpoints are (1) the mean change in 24-hour ambulatory systolic BP from baseline to 12 weeks in patients with hypertension [Category 1 & 3], and (2) the mean change in serum LDL-cholesterol from baseline to 12 weeks in patients with hyperlipidemia [Category 2 & 3].

ELIGIBILITY:
Inclusion Criteria:

* health insurance subscribers who are aged 20-54 years
* 24-hour ambulatory systolic BP 130-159 mmHg or serum LDL ≥130 mg/dl
* Android smartphone users who can use ICT-based helathcare application
* no use of anti-hypertensive or lipid-lowering drugs for ≥3 months prior to screening
* subjects who are considered appropriate to be managed with lifestyle modification for 12 weeks
* Subject who understands the purpose of the study and signs with informed consent form

Exclusion Criteria:

* 24-hour ambulatory systolic or diastolic BP >160 mmHg or > 110 mmHg
* underlying cardiovascular disease (ischemic heart disease, heart failure, aortic disease, valvular heart disease, arrhythmia, cardiomyopathy, etc.)
* underlying cerebrovascular disease (stroke, cerebral infarction or hemorrhage, cerebral aneurysm, etc.)
* chronic renal disease
* peripheral vascular disease
* pregnancy
* secondary hypertension
* atrial fibrillation or flutter
* severe bradyarrhythmia
* difficulty in BP measurement by smart watch
* difference in systolic BP measurements from both arms > 10mmHg
* life expectancy < 2 years
* medical conditions that would limit adherence to participation (as confirmed by physicians)

Ages: 20 Years to 54 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 450 (Estimated)
Dates: Start 2023-03-02 (Estimated); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
Mean change in 24-hour ambulatory systolic BP from baseline to 12 weeks | at 12-week follow-up
  in patients with hypertension [Category 1 & 3]
Mean change in serum LDL-cholesterol level from baseline to 12 weeks | at 12-week follow-up
  in patients with hyperlipidemia [Category 2 & 3]

SECONDARY OUTCOMES:
Mean change in 24-hour ambulatory diastolic BP from baseline to 12 weeks | at 12-week follow-up
Mean change in daytime systolic BP from baseline to 12 weeks | at 12-week follow-up
Mean change in daytime diastolic BP from baseline to 12 weeks | at 12-week follow-up
Mean change in nighttime systolic BP from baseline to 12 weeks | at 12-week follow-up
Mean change in nighttime diastolic BP from baseline to 12 weeks | at 12-week follow-up
change in diurnal variability of BP from baseline to 12 weeks | at 12-week follow-up
percent of subjects achieving the target BP | at 12-week follow-up
percent of subjects achieving the target LDL-cholesterol | at 12-week follow-up
change in serum triglyceride from baseline to 12 weeks | at 12-week follow-up
change in serum HDL-cholesterol from baseline to 12 weeks | at 12-week follow-up
change in body mass index from baseline to 12 weeks | at 12-week follow-up
change in quality of life (EuroQOL) from baseline to 12 weeks | at 12-week follow-up
change in activity score (IPAQ) from baseline to 12 weeks | at 12-week follow-up
change in smart watch-measured mean systolic BP from baseline to 12 weeks | at 12-week follow-up
change in smart watch-measured mean diastolic BP from baseline to 12 weeks | at 12-week follow-up

IPD SHARING:
Plan to Share IPD: No